CLINICAL TRIAL: NCT03083860
Title: Evaluation of Migraine Management Mobile App Combined With Electrophysiological Measurements for Identification of Migraine Attack Risk and Beneficial Preventive Actions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainmarc Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLD10
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: 2 groups of 15-45 patients will be recruited in parallel and monitored for 4-6 weeks, than they will be followed for 4-6 weeks. They will receive feedback based on diary information and EEG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Other): 15-45 participants will be monitored for 4-6 weeks, using the App in a Closed version followed by 4-6 weeks, using the App in an Open version (A version of the app the generates recommendations of ADL interventions) , with feedback based on diary information and BEI; followed by 4-6 weeks using the App in an Open version, with feedback based on diary information only.
  Interventions: Device: BEI
- Arm II (Other): 15-45 participants will be monitored for 4-6 weeks, using the App in a Closed version followed by 4-6 weeks, using the App in an Open version with feedback based on diary information only followed by 4-6 weeks; followed by 4-6 weeks using the App in an Open version, with feedback based on diary information and BEI. Note the difference between Arm I and Arm II is the order of use of BEI in addition to the diary feedback.
  Interventions: Device: BEI

INTERVENTIONS:
Device: BEI — BrainMARC Ltd. has demonstrated in recent years the ability to extract effective attention markers from averaged ERP waves sampled with a single EEG channel (two electrodes). In addition, BrainMARC has developed a template matching method to extract the attention-related markers at the single-trial level. An index (termed Brain Engagement Index - BEI) can then be generated from a 1-minute, single-channel sample.

SUMMARY:
Evaluation of migraine management mobile app combined with electrophysiological measurements for identification of migraine attack risk and beneficial preventive actions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine by a neurologist.
* Male or Female, aged 18 -50 years.
* Having 3-10 migraine attacks per month.
* Able and willing to comply with all study requirements.
* Having Android based smartphone

Exclusion Criteria:

* Diagnosed with chronic pain, neurological or psychiatric disorders.
* Current or past use of anti-depressants.
* A user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence.
* History of seizures.
* Head injury with consciousness loss in the last three months.
* Diagnosed as ADHD and/or use of Ritalin.
* Hearing disorder and/or known eardrum impairment.
* Having migraine attacks occurring only during the menstruation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of correlation of attention-related electrophysiological changes and patients' migraine dynamics based at-home EEG measurements via mobile phone app. | 12 months
  significant difference between interictal days and treictal days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided